CLINICAL TRIAL: NCT05635838
Title: A Phase 2, Double-Blind, Randomized, Vehicle-Controlled, Efficacy, and Safety Study of Ruxolitinib Cream in Participants With Hidradenitis Suppurativa
Brief Title: Study to Evaluate of the Efficacy and Safety of Ruxolitinib Cream in Participants With Hidradenitis Suppurativa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCB 18424-221
Expanded Access: NCT03147742 (Approved for marketing)
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Results first posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis suppurativa; skin disease; ruxolitinb cream
MeSH Terms: conditions — Hidradenitis Suppurativa; Skin Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to 1 of 2 treatment groups (ruxolitinib 1.5% cream BID or vehicle cream BID).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib Cream (Experimental): Ruxolitinib 1.5% cream BID for 16 weeks of double-blind, vehicle-controlled (DBVC) period followed by ruxolitinb 1.5% cream BID for 16 weeks in an open-label extension.
  Interventions: Drug: Ruxolitinib cream
- Vehicle Cream (Experimental): Vehicle cream BID for 16 weeks of double-blind, vehicle-controlled (DBVC) period followed by ruxolitinb 1.5% cream BID for 16 weeks in an open-label extension.
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: Ruxolitinib cream — Ruxolitinib cream is a topical formulation applied as a thin film to affected areas.
  Other Names: INCB018424 cream
  Arms: Ruxolitinib Cream
Drug: Vehicle cream — Vehicle cream is matching in appearance to ruxolitinib cream and is to be applied in the same manner as ruxolitinib cream.
  Arms: Vehicle Cream

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Ruxolitinib cream in participants with Hidradenitis Suppurativa. This is a randomized 16-week double-blind, vehicle-controlled (DBVC) study followed by a 16 week open label extension period (OLE) with an active treatment for participants who complete the DBVC period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HS based on clinical history and physical examination for at least 3 months.
* Diagnosis of HS (Hurley I or II) with the following:

  1. A total AN count of 3 to ≤ 10, with no draining tunnels at screening and baseline visits. AND
  2. The AN count at the screening AND baseline visits:
* AN of 3 should affect at least 1 distinct anatomical area
* AN of > 3 to ≤ 10 should affect at least 2 distinct anatomical areas.
* Baseline Skin Pain or Itch NRS score ≥ 1.
* Agreement to NOT use topical and systemic antibiotics for treatment of HS during the study.
* Agreement to NOT use a diluted beach bath or topical antiseptic washes containing chlorhexidine gluconate or benzoyl peroxide on the areas affected by HS lesions during the study.
* Willingness to avoid pregnancy or fathering children

Exclusion Criteria:

* Presence of draining tunnels at screening or at baseline visits.
* Concurrent conditions and history of other diseases:

  1. Active ongoing inflammatory diseases of the skin other than HS that might confound the evaluation of HS.
  2. Any other concomitant skin disorder (eg, generalized erythroderma such as Netherton's syndrome), pigmentation, or extensive scarring that in the opinion of the investigator may interfere with the evaluation of HS AN or compromise participant safety.
  3. Immunocompromised (eg, lymphoma, acquired immunodeficiency syndrome, or Wiskott-Aldrich syndrome).
  4. Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before baseline.
  5. Active acute bacterial, fungal, or viral skin infection (eg, herpes simplex, herpes zoster, chicken pox, clinically infected AD, or impetigo) within 2 weeks before baseline.
* Laboratory values outside of the protocol-defined criteria.
* Use of any prohibited medications per protocol-defined criteria.
* Pregnant or lactating participants, or those considering pregnancy during the period of their study participation.
* Other exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2024-03-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (15):
  - Medical Dermatology Specialists Phoenix, Phoenix, Arizona
  - First Oc Dermatology, Fountain Valley, California
  - Skin Care Research, Llc Scr Hollywood, Boca Raton, Florida
  - Forcare Clinical Research, Tampa, Florida
  - Marietta Dermatology the Skin Cancer Center Marietta, Marietta, Georgia
  - Delricht Research, Baton Rouge, Louisiana
  - Delricht Research, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Revival Research Institute, Llc Troy, Troy, Michigan
  - Dr Bobby Buka, Md Greenwich Village, New York, New York
  - Dermatology Associates of Plymouth Meeting, Plymouth Meeting, Pennsylvania
  - International Clinical Research Tennessee Llc, Murfreesboro, Tennessee
  - Austin Institute For Clinical Research Aicr Pflugerville, Pflugerville, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Dermatology Specialists of Spokane, Spokane, Washington
- Canada (5):
  - Wiseman Dermatology Research Inc, Winnipeg, Manitoba
  - Dr.Wei Jing Loo Medicine Professional Corp, London, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - Skin Centre For Dermatology, Peterborough, Ontario
  - Xlr8 Medical Research, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 19 study centers in Canada and the United States.
Groups:
- Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID: Participants applied ruxolitinib 1.5% cream twice daily (BID) for 16 weeks.
- DBVC Period: Vehicle Cream BID: Participants applied matching vehicle cream BID for 16 weeks.
- Open-label Extension (OLE) Period: Ruxolitinib 1.5% Cream BID: Participants who completed the Week 16 assessments with no safety concerns could continue into the 16-week OLE Period. Participants who applied ruxolitinib 1.5% cream BID during the DBVC Period continued to apply ruxolitinib 1.5% cream BID for an additional 16 weeks in the OLE Period.
- OLE Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID: Participants who completed the Week 16 assessments with no safety concerns could continue into the 16-week OLE Period. Participants who applied vehicle cream BID during the DBVC Period applied ruxolitinib 1.5% cream BID for 16 weeks in the OLE Period.
Period: 16-Week DBVC Period
Arm/Group | Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID | DBVC Period: Vehicle Cream BID | Open-label Extension (OLE) Period: Ruxolitinib 1.5% Cream BID | OLE Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID
Started | 34 | 35 | 0 | 0
Completed | 24 | 32 | 0 | 0
Not Completed | 10 | 3 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Presence of Disease Tunnel | 1 | 0 | 0 | 0
Not completed — Developed Draining Fistula | 0 | 1 | 0 | 0
Period: 16-Week OLE Period
Arm/Group | Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID | DBVC Period: Vehicle Cream BID | Open-label Extension (OLE) Period: Ruxolitinib 1.5% Cream BID | OLE Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID
Started | 0 | 0 | 24 | 32
Completed | 0 | 0 | 21 | 24
Not Completed | 0 | 0 | 3 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID | DBVC Period: Vehicle Cream BID | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (9.83) | 31.3 (9.84) | 31.7 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 33 | 62
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 1 | 8
  Not Hispanic or Latino | 27 | 34 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 19 | 12 | 31
  Black/African-American | 11 | 18 | 29
  Asian | 0 | 2 | 2
  Unknown | 1 | 0 | 1
  Mixed Race: Black and White | 1 | 0 | 1
  White and American Indian/Alaska Native | 2 | 0 | 2
  Half White, Half Asian | 0 | 1 | 1
  Metis, White | 0 | 1 | 1
  North African | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Abscess and Inflammatory Nodule (AN) Count at Week 16
Description: The mixed model repeated measure (MMRM) included the fixed effects of the treatment group (ruxolitinib 1.5% and vehicle cream), stratification factor (Baseline AN count of ≥3 to 4 or ≥5 to 10), visit, and visit-by-treatment interaction. Change from Baseline was calculated as the Week 16 value minus the Baseline value.
Time Frame: Baseline; Week 16
Population: Intent-to-Treat (ITT) Population: all randomized participants. Treatment groups were defined according to treatment assignment at randomization. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: ANs
Arm/Group | Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 24 | 32
ANs | -3.61 (0.378) | -2.42 (0.336)
Statistical Analysis 1: Comparison: Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID vs DBVC Period: Vehicle Cream BID; Test type: Superiority — Response Variable = Treatment + Baseline AN Count Category (≥3 to 4, ≥5 to 10) + Visit + Treatment*Visit; p = 0.0215, ANCOVA; least squares mean difference = -1.20, 95% CI 2-sided [-2.21 to -0.18], Standard Error of Mean 0.506

2. Secondary Outcome: Percentage of Participants Achieving AN50, AN75, AN90, and AN100 at Week 16
Description: AN50, AN75, AN90, and AN100 were defined as at least a 50%, 75%, 90%, and 100% decrease, respectively, in AN count relative to Baseline.
Time Frame: Baseline; Week 16
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 24 | 32
percentage of participants
  AN50 | 79.2 | 56.3
  AN75 | 54.2 | 25.0
  AN90 | 20.8 | 12.5
  AN100 | 20.8 | 12.5

3. Secondary Outcome: Change From Baseline to Week 16 in Total AN Count in Anatomical Areas With Pre-existing ANs at Baseline
Description: Pre-existing ANs at Baseline were defined as abscesses and/or inflammatory nodules present at Baseline. All new ANs identified during the study in an anatomical area that had pre-existing ANs at Baseline were counted. Any new ANs identified in an anatomical area that was initially free of ANs at Baseline were not counted. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The MMRM included the fixed effects of the treatment group (ruxolitinib 1.5% and vehicle cream), stratification factor (Baseline AN count of ≥3 to 4 or ≥5 to 10), visit, and visit-by-treatment interaction. Change from Baseline was calculated as the Week 16 value minus the Baseline value.
Time Frame: Baseline; Week 16
Population: ITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: ANs
Arm/Group | Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 24 | 32
ANs | -3.85 (0.362) | -3.17 (0.323)
Statistical Analysis 1: Comparison: Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID vs DBVC Period: Vehicle Cream BID; Test type: Superiority — Response Variable = Treatment + Baseline AN Count Category (≥3 to 4, ≥5 to 10) + Visit + Treatment*Visit; p = 0.1671, ANCOVA; least squares mean difference = -0.68, 95% CI 2-sided [-1.65 to 0.29], Standard Error of Mean 0.485

4. Secondary Outcome: Change From Baseline in Skin Pain Numeric Rating Scale (NRS) Score at Week 16
Description: The Skin Pain NRS is a daily participant-reported measure (24-hour recall) of the worst level of skin pain related to Hidradenitis Suppurativa. The participants rated the pain severity of their Hidradenitis Suppurativa by selecting a number from 0 (no pain) to 10 (worst imaginable pain) that best described their worst level of pain in the past 24 hours. The MMRM included the fixed effects of the treatment group (ruxolitinib 1.5% and vehicle cream), stratification factor (Baseline AN count of ≥3 to 4 or ≥5 to 10), visit, and visit-by-treatment interaction. Change from Baseline was calculated as the Week 16 value minus the Baseline value.
Time Frame: Baseline; Week 16
Population: ITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 23 | 22
scores on a scale | -1.90 (0.532) | -2.09 (0.497)
Statistical Analysis 1: Comparison: Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID vs DBVC Period: Vehicle Cream BID; Test type: Superiority — Response Variable = Treatment + Baseline AN Count Category (≥3 to 4, ≥5 to 10) + Visit + Treatment*Visit; p = 0.7982, ANCOVA; least squares mean difference = 0.19, 95% CI 2-sided [-1.27 to 1.64], Standard Error of Mean 0.728

5. Secondary Outcome: Change From Baseline in Itch NRS Score at Week 16
Description: The Itch NRS is a daily participant-reported measure (24-hour recall) of the worst level of itch intensity related to Hidradenitis Suppurativa. The participants rated the itch severity of their Hidradenitis Suppurativa by selecting a number from 0 (no itch) to 10 (worst imaginable itch) that best described their worst level of itching in the past 24 hours. The MMRM included the fixed effects of the treatment group (ruxolitinib 1.5% and vehicle cream), stratification factor (Baseline AN count of ≥3 to 4 or ≥5 to 10), visit, and visit-by-treatment interaction. Change from Baseline was calculated as the Week 16 value minus the Baseline value.
Time Frame: Baseline; Week 16
Population: ITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 23 | 22
scores on a scale | -1.45 (0.538) | -2.39 (0.493)
Statistical Analysis 1: Comparison: Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID vs DBVC Period: Vehicle Cream BID; Test type: Superiority — Response Variable = Treatment + Baseline AN Count Category (≥3 to 4, ≥5 to 10) + Visit + Treatment*Visit; p = 0.2031, ANCOVA; least squares mean difference = 0.94, 95% CI 2-sided [-0.52 to 2.40], Standard Error of Mean 0.730

6. Secondary Outcome: Percentage of Participants Who Achieve Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 16
Description: HiSCR was defined as at least a 50% reduction in AN count with no increase in either abscess or draining fistula counts, relative to Baseline.
Time Frame: Baseline; Week 16
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 24 | 32
percentage of participants | 79.2 | 50.0

7. Secondary Outcome: Change From Baseline in the International Hidradenitis Suppurativa Severity Score System (IHS4) Score at Week 16
Description: The IHS4 is a composite, dynamic score and validated tool used to determine Hidradenitis Suppurativa severity. IHS4 score was calculated by the number of inflammatory nodules (multiplied by 1) plus the number of abscesses (multiplied by 2) plus the number of draining tunnels (multiplied by 4). Scores: mild=0-3; moderate=4-10; severe ≥11. The MMRM included the fixed effects of the treatment group (ruxolitinib 1.5% and vehicle cream), stratification factor (Baseline AN count of ≥3 to 4 or ≥5 to 10), visit, and visit-by-treatment interaction. Change from Baseline was calculated as the Week 16 value minus the Baseline value.
Time Frame: Baseline; Week 16
Population: ITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 24 | 32
scores on a scale | -3.58 (0.505) | -2.76 (0.459)
Statistical Analysis 1: Comparison: Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID vs DBVC Period: Vehicle Cream BID; Test type: Superiority — Response Variable = Treatment + Baseline AN Count Category (≥3 to 4, ≥5 to 10) + Visit + Treatment*Visit; p = 0.2387, ANCOVA; least squares mean difference = -0.82, 95% CI 2-sided [-2.20 to 0.56], Standard Error of Mean 0.683

8. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE ) in the Double-blind, Vehicle-controlled (DBVC) Period
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. A TEAE was defined as any AE reported for the first time or the worsening of a pre-existing event after the first application of study drug.
Time Frame: up to Week 16 plus 30 days
Population: Safety Population: all participants who applied ruxolitinib 1.5% cream or vehicle cream at least once. Treatment groups were determined according to the actual treatment the participant applied on Day 1 regardless of assigned treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 34 | 35
Participants | 13 | 15

9. Secondary Outcome: Number of Participants With Any Grade 3 or Higher TEAE in the DBVC Period
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. A TEAE was defined as any AE reported for the first time or the worsening of a pre-existing event after the first application of study drug. The severity of AEs was assessed using Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grades 1 through 5. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: up to Week 16 plus 30 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 34 | 35
Participants | 0 | 2

10. Secondary Outcome: Number of Participants With Any TEAE in the Open-label Extension (OLE) Period
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. A TEAE was defined as any AE reported for the first time or the worsening of a pre-existing event after the first application of study drug.
Time Frame: from Week 17 up to Week 32 plus 30 days
Population: Open-label Extension Safety Population: all participants who applied ruxolitinib 1.5% cream BID at least once during the OLE Period
Measure: Count of Participants; unit: Participants
Groups:
- OLE Period: Ruxolitinib 1.5% Cream BID: Participants who completed the Week 16 assessments with no safety concerns could continue into the 16-week OLE Period. Participants who applied ruxolitinib 1.5% cream BID during the DBVC Period continued to apply ruxolitinib 1.5% cream BID for an additional 16 weeks in the OLE Period.
Arm/Group | OLE Period: Ruxolitinib 1.5% Cream BID | OLE Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 24 | 32
Participants | 8 | 15

11. Secondary Outcome: Number of Participants With Any Grade 3 or Higher TEAE in the OLE Period
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. A TEAE was defined as any AE reported for the first time or the worsening of a pre-existing event after the first application of study drug. The severity of AEs was assessed using CTCAE v5.0 Grades 1 through 5. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: from Week 17 up to Week 32 plus 30 days
Population: Open-label Extension Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Ruxolitinib 1.5% Cream BID | OLE Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 24 | 32
Participants | 0 | 3

ADVERSE EVENTS:
Time Frame: up to Week 32 plus 30 days
Description: Treatment-emergent adverse events, defined as adverse events reported for the first time or the worsening of pre-existing events after the first application of study drug, have been reported. For safety analysis, participants who transitioned from treatment with vehicle cream BID to treatment with ruxolitinib 1.5% cream BID in the Open-label Extension Period have been counted both in the vehicle arm and the ruxolitinib arm.
Groups:
- Vehicle Cream BID: Participants applied matching vehicle cream twice a day (BID) for 16 weeks in the Double-blind, Vehicle-controlled Period.
- Ruxolitinib 1.5% Cream BID: Participants applied ruxolitinib 1.5% cream BID during the Double-blind, Vehicle-controlled (DBVC) Period and the Open-label Extension (OLE) Period. Participants applied ruxolitinib 1.5% cream BID for 16 weeks in the DBVC Period. Participants who completed the Week 16 assessments with no safety concerns could continue into the 16-week OLE Period. Participants who applied ruxolitinib 1.5% cream BID during the DBVC Period continued to apply ruxolitinib 1.5% cream BID for an gadditional 16 weeks in the OLE Period. Participants who applied vehicle cream BID during the DBVC Period applied ruxolitinib 1.5% cream BID for 16 weeks in the OLE Period.
Arm/Group | Vehicle Cream BID | Ruxolitinib 1.5% Cream BID
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/66
Serious Adverse Events (participants affected / at risk) | 1/35 | 2/66
Other Adverse Events (participants affected / at risk) | 2/35 | 5/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Cream BID (N=35) | Ruxolitinib 1.5% Cream BID (N=66)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Cream BID (N=35) | Ruxolitinib 1.5% Cream BID (N=66)
Nasopharyngitis (Infections and infestations) | 0 (0) | 5 (5)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT05635838/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT05635838/SAP_001.pdf